CLINICAL TRIAL: NCT05009810
Title: Efficacy and Safety of Astaxanthin in Volunteer With Refraction Errors
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Chulalongkorn University (Other)
Responsible Party: Principal Investigator, Pornanong Aramwit, Pharm.D., Ph.D, Professor, Chulalongkorn University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: EC2103320
Record Dates: First submitted 2021-08-03; First posted 2021-08-18 (Actual); Last update posted 2021-08-18 (Actual); Status verified 2021-08

CONDITIONS: Refractive Errors
MeSH Terms: conditions — Refractive Errors | interventions — astaxanthine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- astaxanthin 4 mg (Experimental): The astaxanthin 4 mg will be taken 1 capsule once daily for 2 months.
  Interventions: Dietary Supplement: astaxanthin 4 mg
- astaxanthin 6 mg (Experimental): The astaxanthin 6 mg will be taken 1 capsule once daily for 2 months.
  Interventions: Dietary Supplement: astaxanthin 6 mg
- Placebo (Placebo Comparator): The placebo will be taken 1 capsule once daily for 2 months.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: astaxanthin 4 mg — They will take astaxanthin 4 mg 1 capsule once daily for 2 months.
  Arms: astaxanthin 4 mg
Dietary Supplement: astaxanthin 6 mg — They will take astaxanthin 6 mg 1 capsule once daily for 2 months.
  Arms: astaxanthin 6 mg
Dietary Supplement: Placebo — They will take placebo 1 capsule once daily for 2 months.
  Arms: Placebo

SUMMARY:
This study will investigate efficacy and safety of astaxanthin in 180 volunteers with refraction errors. Visual test, skin test, liver function test, renal function test, and adverse event will be evaluated before and after taking astaxanthin for 1 and 2 months.

DETAILED DESCRIPTION:
This study will investigate efficacy and safety of astaxanthin in 180 volunteers with refraction errors. They will divided into 3 groups which are astaxanthin 4 mg group , astaxanthin 6 mg group, and placebo group. They will take the sample 1 capsule once daily for 2 months. Visual test, skin test, liver function test, renal function test, and adverse event will be evaluated before and after taking the sample for 1 and 2 months.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-65 years
* Refraction errors, dry eye, or blurred vision
* Have a willingness to participate in the study

Exclusion Criteria:

* Uncontrolled disease
* Have complications during the study
* Have astaxanthin more than 2 weeks
* Allergic to astaxanthin, seafood, or seaweed
* Osteoporosis or thyroid disease
* Immunodeficiency or taking immunosuppressants
* Liver and kidney diseases
* A person with a brain disorder, vision or hearing unusual
* Pregnancy or lactation
* Cannot follow the protocol
* During participated in other studies

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2021-08-15 (Estimated); Primary Completion 2022-06-30 (Estimated); Study Completion 2022-07-31 (Estimated)

PRIMARY OUTCOMES:
Visual acuity value | 2 months
  Measured using Snellen Chart (logarithm of the minimal angle of resolution unit)

SECONDARY OUTCOMES:
Refractive status | 2 months
  Measured using Auto refractometer (two digit scale)
Eye fatigue status | 2 months
  Measured using eye fatigue questionnaire (scale 1 to 5 which are no symptom (1) to severe(5))
Vision status | 2 months
  Measured using Thai National Eye Institute Visual Functioning Questionnaire 25 (scale 25 to 100 which are normal (25) to worse(100))
Skin erythema value | 2 months
  Measured using Mexameter (skin erythema index)
Skin melanin value | 2 months
  Measured using Mexameter (skin melanin index)
Skin humidity value | 2 months
  Measured using Corneometer (skin humidity index)
Skin transepidermal water loss value | 2 months
  Measured using Transepidermal water loss meter (skin transepidermal water loss index)
Aspartate transaminase value | 2 months
  Measured aspartate transaminase value (U/L) in blood
Alanine aminotransferase value | 2 months
  Measured alanine aminotransferase value (U/L) in blood
Alkaline phosphatase value | 2 months
  Measured alkaline phosphatase value (U/L) in blood
Blood urea nitrogen value | 2 months
  Measured blood urea nitrogen value (mg/dl) in blood
Creatinine value | 2 months
  Measured creatinine value (mg/dl) in blood
Adverse events | 2 months
  Measured using questionnaire (Yes or No)